CLINICAL TRIAL: NCT05879692
Title: Response of Irritable Bowel Syndrome to Abdominal Fat Reduction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aly Elrashidy, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/004475
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Irritable Bowel Syndrome; Obesity; Abdominal Obesity
Keywords: Irritable Bowel Syndrome; abdominal fat; central obesity; high intensity focused ultrasound; FODMAPs diet
MeSH Terms: conditions — Irritable Bowel Syndrome; Obesity; Obesity, Abdominal | interventions — Caloric Restriction; Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Group A) (Experimental): Will consist of 30 cases suffering from mild to moderate Irritable Bowel Syndrome (IBS) with mild to moderate obesity will receive High Intensity Focused Ultrasound (Cavitation), a dietary regimen that combines Low Caloric Diet (LCD) and low (FODMAPs) diet and aerobic exercises with moderate intensity.
  Interventions: Procedure: focused ultrasound; Behavioral: Low Caloric Diet (LCD) and a low (FODMAPs) diet; Other: aerobic exercise
- control group (Group B) (Active Comparator): Will consist of 30 cases suffering from mild to moderate Irritable Bowel Syndrome (IBS) with mild to moderate obesity will receive only the same dietary regimen and aerobic exercise that prescribed for group A.
  Interventions: Behavioral: Low Caloric Diet (LCD) and a low (FODMAPs) diet; Other: aerobic exercise

INTERVENTIONS:
Procedure: focused ultrasound — focused ultra sound cavitation using a device of Mabel6 DUO Ultra Cavitation Technology system produced by DAEYANG MEDICAL COMPANY, KOREA will be applied on the abdominal region which extending bilaterally from the line extending from mid axilla to iliac crest, and above from center of diaphragm to the line extending between two iliac crest below.
  the session of Focused Ultra Sound will take 25- 30 minutes, twice/week and with about three day intervals for 12 weeks.
  Other Names: cavitation
  Arms: study group (Group A)
Behavioral: Low Caloric Diet (LCD) and a low (FODMAPs) diet — The Low caloric diet (LCD) diet will be an equilibrated diet that had a caloric value 10% below the total metabolic expenditure (total energy expenditure) of each individual.
  The low FODMAPs diet (LFD) is a diet low in fermentable oligo-, di-, mono- saccharides and polyols (FODMAPs).
  Other Names: dietary regimen
Other: aerobic exercise — aerobic exercise program under direct supervision at a frequency of 3 times/week for 12 weeks, in the form of walking on a treadmill for 30 minutes with moderate intensity (12-14) according to The Borg Rating of Perceived Exertion (RPE) scale.

SUMMARY:
The purpose of the study is to find out the response of Irritable Bowel Syndrome (IBS) to abdominal fat reduction in central obese patients using: application of High Intensity Focused Ultrasound (cavitation) on the abdominal region, aerobic exercise and a dietary regimen that will be low in calories (Low Caloric Diet) and low in fermentable oligo-, di-, mono- saccharides and polyols (low-FODMAPs).

DETAILED DESCRIPTION:
Irritable bowel syndrome is a common functional gastrointestinal (GI) disorder, with a high global prevalence and a strong impact on the quality of life. There is a positive association between irritable bowel syndrome (IBS) and increased BMI and volume of android fat, according to waist circumference.

Central obesity and Irritable Bowel Syndrome (IBS) are common medical conditions with similar etiologic mechanisms. There are several studies considering obesity as the risk factor for (IBS), but limited studies that to evaluate the association between abdominal obesity and the incidence of irritable bowel syndrome (IBS). Establishing such association is important in the management of IBS.

Focused ultra sound cavitation is a noninvasive safe technique for reducing localized subcutaneous adipose tissue by generating molecular vibrations that elevate the local tissue temperature and produce rapid cell necrosis in targeted tissues.

the investigators believe that focused ultrasound cavitation could improve the overall of Irritable Bowel Syndrome severity as a consequence of abdominal fat reduction.

To the best of the investigators' knowledge, there are limited studies to confirm the improvement of irritable bowel syndrome (IBS) as a result of abdominal fat reduction by focused ultrasound cavitation.

Therefore, this study is a trial to investigate the effect of focused ultrasound cavitation augmented with aerobic exercise and dietary regimen on improvement of Irritable bowel syndrome (IBS) in patients with central obesity.

Sixty volunteer central obese patients (males and females) with Irritable Bowel Syndrome (IBS) which will be diagnosed according to Rome IV criteria will be participated in this study and will be referred from the Gastroenterology outpatient clinic of El-Sahel Teaching Hospital, Cairo. The study will be conducted at El-Sahel Teaching Hospital.

ELIGIBILITY:
Inclusion Criteria:

* All patients will be 20-45 years of age.
* Both genders will be participated.
* sedentary (exercise < 2 times/week).
* Body mass index (BMI) will be ranged from 30 to 39.9 kg/m² and their waist circumference ≥ 102 cm for men and ≥ 88 cm for women.
* Patients will have the criteria of Irritable Bowel Syndrome (IBS) according to Rome IV Which are: recurrent abdominal pain on average at least one day per week during the previous three months associated with two or more of the following features must fulfill: (1) Pain is related to defecation; (2) Pain associated with a change in frequency of stool; and (3) Pain associated with a change in form or appearance of stool.
* mild to moderate Irritable Bowel Syndrome with score of 75- 300 according to the questionnaire of Irritable Bowel Syndrome Severity Scoring System (IBS-SSS).

Exclusion Criteria:

* • Under 20 or above 45 years of age.

  * Athletics
  * Musculoskeletal, Carcinogenic, or kidney diseases, diabetes, hepatitis and cardiac disorders.
  * Any condition that may prevent the use of the focused ultrasound on the abdominal region such as scarring, hernias or skin diseases in the abdominal area.
  * Patients with severe Irritable Bowel Syndrome (IBS) or other known organic gastrointestinal disorders rather than IBS including: (1) Fever, Weight loss or Jaundice; (2) Change in the color of stool; (3) Signs of anemia or Thyroid disease; (4) Abdominal mass or Organomegaly; (5) Signs of intestinal obstruction.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-28 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
change in total body fat percentage | change from baseline total body fat percentage at 12 weeks
  total body fat percentage will be measured by Dual-energy X-ray Absorptiometry (DXA)
change in abdominal subcutaneous fat percentage | change from baseline abdominal subcutaneous fat percentage at 12 weeks
  abdominal subcutaneous fat percentage will be measured by Dual-energy X-ray Absorptiometry (DXA)
change in abdominal visceral fat percentage | change from baseline abdominal visceral fat percentage at 12 weeks
  abdominal visceral fat percentage will be measured by Dual-energy X-ray Absorptiometry (DXA)
change in Irritable bowel syndrome Severity Scoring system (IBS-SSS) | change from baseline Irritable bowel syndrome Severity Scoring system at 12 weeks
  The Irritable bowel syndrome Severity Scoring System (IBS-SSS) questionnaire was validated by Francis et al. in 1997and consists of five questions that measure: (1) abdominal pain severity; (2) frequency (number of days in every 10 days) with abdominal pain; (3) abdominal bloating/distension; (4) satisfaction with bowel habits; (5) IBS-related quality of life (QoL). Each measure is rated from 0 to 100, with total scores ranging from 0 to 500
change in Irritable bowel syndrome-quality of life (IBS-QOL) | change from baseline Irritable bowel syndrome-quality of life at 12 weeks
  The Irritable bowel syndrome-quality of life questionnaire (IBS-QOL) consists of 34 items assessing patients' well-being across eight subscales: dysphoria (eight items); interference with activity (seven items); body image (four items); social reaction (four items); health worry (three items); food avoidance (three items); relationships (three items); and sexual (two items)

SECONDARY OUTCOMES:
change in body weight | change from baseline body weight at 12 weeks
  Weight scale will be used to measure the weight (in kilograms) of all patients in both groups (A & B)
change in body mass index | change from baseline body mass index at 12 weeks
  Body Mass Index (BMI) is calculated as body weight (in kilograms) divided by the square of body height (in meters) (BMI= Kg/m²)
change in waist circumference measurement | change from baseline Waist circumference at 12 weeks
  Waist circumference (WC) will be measured (in centimeters) by the tape measurement at the midway between the lowest rib and the iliac crest, while the patient in the standing position with light clothes and at the end of expiration

CONTACTS AND LOCATIONS:
Overall Officials: Aly S Elrashidy, M.Sc., Principal Investigator — Cairo University
Locations (1):
- El-Sahel Teaching Hospital, Cairo, Egypt